CLINICAL TRIAL: NCT04379141
Title: Ultrasonic Measurement of Inferior Vena Cava and Internal Jugular Vein in Predicting Hypotension After Anesthesia Induction in Patients Undergoing Gastrointestinal Surgery
Brief Title: Ultrasonic Measurement of IVC and IJV in Predicting Hypotension After Anesthesia Induction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jin Dong Liu (Other)
Responsible Party: Sponsor-Investigator, Jin Dong Liu, The Affiliated Hospital of Xuzhou Medical University, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Other Study IDs: XYFY2019-1202
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypotension: Patients with hypotension after induction of anesthesia
- non-hypotension: Patients without hypotension after induction of anesthesia

SUMMARY:
This research is expected to study ultrasonic measurement of internal jugular vein and inferior vena cava, which can be used as a good index to predict hypotension after anesthesia induction, and its measurement method is simple and quick.

DETAILED DESCRIPTION:
The induction of anesthesia is the process from the physiological state to the anesthetic state in a short period of time. Hypotension after anesthesia induction is closely related to many organ injuries. Gastrointestinal surgery patients' prohibition of fasting is an important mechanism of severe hypotension after anesthesia induction. At present, ultrasonic measurement of inferior vena cava and internal jugular vein has been proved to be a convenient and non-invasive means to evaluate patients' blood volume. The purpose of this research was to study the relativity between ultrasonic measurement of inferior vena cava and internal jugular vein and hypotension after anesthesia induction in patients.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal surgery
* BMI 18~24
* ASA score gradeⅠ~ III

Exclusion Criteria:

* anemia
* cirrhosis
* Emergency surgery
* severe hypertension
* New York Heart Association III ~ IV or ejection fraction <40%
* cirrhosis
* Other serious systemic diseases

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing gastrointestinal surgery in the Affiliated Hospital of Xuzhou Medical University
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-05-08 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension after anesthesia Induction | within 12 hours after anesthesia induction
  Hypotension can be diagnosed if one of the following conditions is true: (1) a decrease in mean arterial pressure of > 20% compared to the baseline value (2) mean arterial pressure < 60mmHg

SECONDARY OUTCOMES:
Ultrasonic measurement of inferior vena cava and internal jugular vein | within 1 hour before anesthesia induction
  Measure the maximum diameter, minimum diameter and cross-sectional area of inferior vena cava and internal jugular vein

CONTACTS AND LOCATIONS:
Overall Officials: Jin Dong Liu, Study Director — The Affiliated Hospital of Xuzhou Medical University

IPD SHARING:
Plan to Share IPD: No